CLINICAL TRIAL: NCT06370689
Title: Comparison of Three Pre-oxygenation Strategies for Prehospital Anaesthesia Induction in Children, Normal Weight Adults and Obese Adults
Brief Title: Comparison of Three Pre-oxygenation Strategies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Mountain Emergency Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PRE-OX
Record Dates: First submitted 2024-04-11; First posted 2024-04-17 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Emergencies; Anesthesia
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (9):
- NRM - Non-rebreather mask in children 6-12 yrs (Active Comparator): Non-rebreather mask in children 6-12 yrs
  Interventions: Other: Preoxygenation
- BVM with PEEP in children 6-12 yrs (Active Comparator): Bag valve mask with positive end-expiratory pressure (PEEP) in children 6-12 yrs
  Interventions: Other: Preoxygenation
- BVM without PEEP in children 6-12 yrs (Active Comparator): Bag valve mask without positive end-expiratory pressure (PEEP) in children 6-12 yrs
  Interventions: Other: Preoxygenation
- NRM - Non-rebreather mask in normal weight adults (Active Comparator): Non-rebreather mask in normal weight adults
  Interventions: Other: Preoxygenation
- BVM with PEEP in normal weight adults (Active Comparator): Bag valve mask with positive end-expiratory pressure (PEEP) in normal weight adults
  Interventions: Other: Preoxygenation
- BVM without PEEP in normal weight adults (Active Comparator): Bag valve mask without positive end-expiratory pressure (PEEP) in normal weight adults
  Interventions: Other: Preoxygenation
- NRM - Non-rebreather mask in overweight/obese adults (Active Comparator): Non-rebreather mask in overweight/obese adults
  Interventions: Other: Preoxygenation
- BVM with PEEP in overweight/obese adults (Active Comparator): Bag valve mask with positive end-expiratory pressure (PEEP) in overweight/obese adults
  Interventions: Other: Preoxygenation
- BVM without PEEP in overweight/obese adults (Active Comparator): Bag valve mask without positive end-expiratory pressure (PEEP) in overweight/obese adults
  Interventions: Other: Preoxygenation

INTERVENTIONS:
Other: Preoxygenation — Preoxygenation of volunteers over 3 minutes

SUMMARY:
Study objective: Comparing the efficacy of three different preoxygenation strategies, i.e. non-rebreather face mask (NRM), bag-valve-mask (BVM) with and BVM without additional positive end-expiratory pressure (PEEP) in three subgroups of spontaneously breathing volunteers.

Study endpoints

Primary Endpoint:

Difference in expiratory oxygen concentration (FeO2) at the end of the 3 min preoxygenation sessions.

Secondary endpoints:

* Difference in Oxygen Reserve Index (ORi) at the end of the 3 min preoxygenation sessions.
* Changes in regional ventilation from baseline to 1.5 min and 3 min into the preoxygenation sessions, assessed using electrical impedance tomography (EIT)
* Time to reaching an Oxygen Reserve Index (ORi) ≥ 0.5
* Time to reaching an Oxygen Reserve Index (ORi) =1
* Time to Oxygen Reserve Index (ORi) back to baseline after the 3 min preoxygenation sessions.

Number of participants 15 participants per subgroup, i.e. 45 participants in total.

Inclusion criteria

* Normal-weight adults (body mass index, BMI 18.5-24.9 kg/m2) with an "American Society of Anesthesiologists Physical Status Classification System (ASA) " score of I or II
* Adults with a BMI 25-39.9 kg/m2 with and ASA score <3
* Healthy (ASA I) children aged 6-12 years Exclusion criteria ASA 3, Age < 6 and age 12-18, pregnant women, missing informed consent, signs and symptoms of an acute respiratory illness on the study day.

After informed consent and a medical check-up, baseline measurements will be done for 10 minutes (peripheral oxygen saturation SpO2, ORI, regional ventilation). Then the participants will undergo 3 different preoxygenation sessions with the 3 interfaces (i.e. non-rebreather facemask with reservoir and a bag-valve-mask with and without PEEP) in a randomized order and a 20 min washout between the sessions. Each preoxygenation session is conducted in a supine position and will be proceeded until the measured FeO2 (end expiratory O2 fraction) reaches 90% or up to a maximum time of 3 min. Afterwards 10 min of SpO2, ORI and regional ventilation measurements will follow.

ELIGIBILITY:
Inclusion Criteria:

* Normal-weight adults (BMI 18.5-24.9 kg/m2) with an "American Society of Anesthesiologists Physical Status Classification System (ASA) " score of I or II
* Adults with a BMI 25-39.9 kg/m2 with and ASA score <3
* Healthy (ASA I) children aged 6-12 years

Exclusion Criteria:

* ASA 3
* Age < 6 and age 12-18
* pregnant women
* missing informed consent
* signs and symptoms of an acute respiratory illness on the study day

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Difference in expiratory oxygen concentration (FeO2) at the end of the 3 min preoxygenation sessions. | After 3 minutes of preoxygenation
  Difference in expiratory oxygen concentration (FeO2) at the end of the 3 min preoxygenation sessions between the three arms.

SECONDARY OUTCOMES:
Difference in Oxygen Reserve Index (ORi) at the end of the 3 min preoxygenation sessions. | After 3 minutes of preoxygenation
  Difference in Oxygen Reserve Index (ORi) at the end of the 3 min preoxygenation sessions. ORi ranges from 0.0 to 1.0 and reflects the partial pressure of oxygen in arterial blood (PaO2 80-200).
Changes in regional ventilation from baseline to 1.5 min and 3 min into the preoxygenation sessions, assessed using electrical impedance tomography (EIT) | After 1.5 and 3 minutes of preoxygenation
  Changes in regional ventilation from baseline to 1.5 min and 3 min into the preoxygenation sessions, assessed using electrical impedance tomography (EIT)
Time to reaching an Oxygen Reserve Index (ORi) ≥ 0.5 | Variable, timepoint during the 3 min preoxygenation session
  Time to reaching an Oxygen Reserve Index (ORi) ≥ 0.5
Time to reaching an Oxygen Reserve Index (ORi) =1 | Variable, timepoint during the 3 min preoxygenation session
  Time to reaching an Oxygen Reserve Index (ORi) =1
Time to Oxygen Reserve Index (ORi) back to baseline after the 3 min preoxygenation sessions. | Washout phase after the 3 min preoxygenation sessions.
  Time to Oxygen Reserve Index (ORi) back to baseline after the 3 min preoxygenation sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Rauch, MD, PhD, Principal Investigator — Institute of Mountain Emergency Medicine, Eurac Research
Locations (1):
- TerraXCube, Bolzano, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roveri G, Camporesi A, Hofer A, Kahlen S, Breidt F, Rauch S. Preoxygenation With and Without Positive End-Expiratory Pressure in Lung-Healthy Volunteers: A Randomized Clinical Trial. JAMA Netw Open. 2025 May 1;8(5):e2511569. doi: 10.1001/jamanetworkopen.2025.11569. PMID 40392551